CLINICAL TRIAL: NCT03693157
Title: The Safety and Efficacy of Current FFR Measurement in NTUH Health Care System
Brief Title: The Safety and Efficacy of FFR Protocol in NTUH System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Other Study IDs: 107-052-E
Record Dates: First submitted 2018-09-27; First posted 2018-10-02 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Bradyarrhythmia; Dyspnea; Acute Respiratory Failure
MeSH Terms: conditions — Bradycardia; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
FFR-guided PCI has been performed in National Taiwan University Hospital(NTUH) for many years. Nevertheless, the method of FFR measurement in NTUH is different from that in literature. In this study, the investigator would like to evaluate the effectiveness and safety of NTUH experience in FFR prospectively. First, the investigator will record any intracoronary (IC) injected adenosine-related complications, such as bradyarrhythmia or chest discomfort. Second, the investigator will follow up on the clinical outcome of the participants for 2 years, record if any target lesion failure, target vessel failure, target vessel-related myocardial infarction, and cardiac death. Finally, left ventricular diastolic pressure, serum pro-brain natriuretic peptide (pro-BNP), and high sensitivity C- reactive protein (hsCRP) will be checked and determined their relationships with the maximum dosage of IC adenosine.

DETAILED DESCRIPTION:
FFR has been introduced for the determination of physiological ischemia in the myocardium for many years. Nowadays, FFR-guided PCI is highly recommended for the assessment of physiologic ischemia in intermediate coronary lesions. FFR-guided PCI has been performed in National Taiwan University Hospital(NTUH) for many years. Nevertheless, the method of FFR measurement in NTUH is different from that in literature. In this study, the investigator would like to evaluate the effectiveness and safety of NTUH experience in FFR prospectively. First, the investigator will record any intracoronary (IC) injected adenosine-related complications, such as bradyarrhythmia or chest discomfort. Second, the investigator will follow up on the clinical outcome of the participants for 2 years, record if any target lesion failure, target vessel failure, target vessel-related myocardial infarction, and cardiac death. Finally, left ventricular diastolic pressure, serum pro-brain natriuretic peptide (pro-BNP), and high sensitivity C- reactive protein (hsCRP) will be checked and determined their relationships with the maximum dosage of IC adenosine.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for FFR examination

Exclusion Criteria:

* Hypersensitivity to adenosine
* Severe valvular aortic stenosis
* Resting heart rate less than 50 beats per minute

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who had intermediate lesion over the coronary artery and eligible for FFR examination
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-11-07 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Adenosine related adverse event | 24 hours
  Including
  1. Bradyarrhythmia including sinus pause and transient AV block
  2. Acute respiratory failure define by respiratory distress which need mechanical ventilator support
Major adverse cardiac event (MACE) | 2 year
  MACE including target lesion failure, target vessel failure, target vessel-related myocardial infarction, and cardiac death

SECONDARY OUTCOMES:
The relationship between left ventricular diastolic pressure and maximum dosage of IC adenosine | 1 hour
  Determine the correlation of left ventricular diastolic pressure and peak dosage of IC adenosine with FFR protocol in NTUH system

OTHER OUTCOMES:
The relationship between pro-BNP,hs-CRP and maximum dosage of IC adenosine | 1 day
  Determine the correlation of pro-BNP,,hs-CRP and peak dosage of IC adenosine with FFR protocol in NTUH system

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Boon Jong, MD, Principal Investigator — National Taiwan University Hospital, Hsinchu Branch.
Locations (1):
- National Taiwan University Hospital Hsin-Chu branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided